CLINICAL TRIAL: NCT03660345
Title: Pars Plana Vitrectomy With Internal Limiting Membrane Peeling Versus Intravitreal Ziv-Aflibercept for Treatment-Naïve Diabetic Macular Edema
Brief Title: PPV With Internal Limiting Membrane Peeling for Treatment-Naïve DME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rush Eye Associates (Other)
Responsible Party: Principal Investigator, Sloan W. Rush, MD, Physician, Rush Eye Associates
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Retina 1
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Diabetic Retinopathy; Macular Edema
MeSH Terms: conditions — Diabetic Retinopathy; Macular Edema | interventions — Intravitreal Injections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPV/MP (Experimental): Study Group: Treatment-naïve subjects with center-involved diabetic macular edema undergo pars plana vitrectomy with internal limiting membrane peeling
  Interventions: Procedure: PPV/MP
- Intravitreal Injection (Active Comparator): Control Group: Treatment-naïve subjects with center-involved diabetic macular edema undergo intravitreal ziv-aflibercept monotherapy according to a fixed treatment schedule
  Interventions: Drug: Intravitreal injection

INTERVENTIONS:
Procedure: PPV/MP — 23 gauge Pars Plana Vitrectomy with Internal Limiting Membrane Peeling
  Arms: PPV/MP
Drug: Intravitreal injection — Intravitreal ziv-Aflibercept
  Arms: Intravitreal Injection

SUMMARY:
Treatment-naïve subjects with center-involved diabetic macular edema undergoing pars plana vitrectomy with internal limiting membrane peeling will have similar visual outcomes but better anatomical outcomes compared to subjects undergoing intravitreal bevacizumab monotherapy at one year.

DETAILED DESCRIPTION:
Diabetic retinopathy is the number one cause of vision loss in working-age adults, and macular edema is the most frequent cause of visual impairment in diabetic patients. Diabetic macular edema (DME) has been treated by a number of different modalities including focal and grid laser, intravitreal corticosteroids, intravitreal anti-vascular endothelial growth factor (VEGF) medications, and pars plana vitrectomy (PPV) with or without internal limiting membrane peeling.

PPV for the treatment of DME was first described in 1992 by Lewis et al, and since then has been studied by numerous investigators under a variety of different clinical settings including the presence of epiretinal membranes, vitreomacular traction (VMT), and diffuse DME. The postulated mechanisms by which PPV may improve DME have included a reduction in macular tangential and anterior-posterior traction, improved oxygenation of the vitreous cavity, and enhanced diffusion of vasogenic growth factors. Other factors that may modulate the response to PPV comprise the patient's lens status and the presence of macular ischemia.

PPV for DME has usually been considered only in patients that responded poorly to other interventions such as laser and/or intravitreal therapy. Typically, such patients have chronic and diffuse DME with, or without, concomitant VMT. Several small prospective, controlled trials have been performed to assess the merits of PPV as a treatment option for such recalcitrant cases with generally disappointing functional outcomes despite having structural improvements. However, since PPV was reserved as a last-ditch effort following a long ordeal with what included multiple lasers and/or intravitreal injections, it should not be surprising that visual outcomes were poor under such circumstances. Presumably most of these patients already would have had irreversible damage to the retina with little or no potential for visual acuity improvement no matter what the intervention might have been. Currently, there are no reports in the literature evaluating PPV as an initial treatment for DME. In this study, we compare PPV to anti-VEGF monotherapy in treatment-naïve subjects with DME in order to evaluate the potential role of PPV in the management of DME before irreversible retinal damage caused by long-standing and persistent DME has set in.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patient able and willing to provide informed consent
3. Diagnosis of diabetes mellitus (type 1 or type 2) is established.
4. Patient has non-proliferative diabetic retinopathy and is treatment-naïve for diabetic retinopathy in the study eye. (Patients may NOT have received treatment of any kind for diabetic retinopathy to the study eye).
5. Best corrected visual acuity letter score is 20/32 or worse, and 20/400 or better at the time of randomization in the study eye.
6. On clinical exam, definite retinal thickening due to diabetic macular edema involving the center of the macula is present in the study eye.
7. Central subfield thickness on the spectral domain OCT is greater than 300 microns at the time of randomization in the study eye.

   (The investigator must verify accuracy of OCT scan by ensuring it is centered and of adequate quality).
8. The study eye has no history of intraocular surgery within the previous four months. Previous uncomplicated cataract surgery otherwise shall be allowed if the study eye is longer than four months out at the time of randomization.

Exclusion Criteria:

1. Proliferative diabetic retinopathy of any kind including neovascularization of the disc/retina/iris, presence of any degree of vitreous hemorrhage, and tractional retinal detachment must be excluded.
2. Patients that received treatment to the posterior segment for any retinal condition must be excluded. Such treatments include intravitreal injections of any kind, retinal lasers of any kind, and subtenons injections.
3. The study eye has a history of previous anterior or pars plana vitrectomy for any reason must be excluded.
4. The patient has a history of systemic anti-VEGF therapy or systemic corticosteroid therapy within the previous 12 months.
5. The patient's macular edema is considered to be due to a cause other than diabetic macular edema.
6. An ocular condition is present such that, in the opinion of the investigator, visual acuity loss would not improve from resolution of macular edema (e.g., foveal atrophy, pigment abnormalities, dense subfoveal hard exudates, a nonretinal condition like corneal scarring or advanced optic nerve cupping from glaucoma, etc.).
7. Substantial cataract that, in the opinion of the investigator, is likely decreasing visual acuity by three or more lines on its own merit (apart from the macular edema).

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
BCVA | 6 months
  Best-corrected visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Sloan Rush, Study Chair — panhandle eye group
Locations (1):
- Hospital La Carlota, Montemorelos, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rush RB, Rush SW. Pars Plana Vitrectomy with Internal Limiting Membrane Peeling for Treatment-Naive Diabetic Macular Edema: A Prospective, Uncontrolled Pilot Study. Clin Ophthalmol. 2021 Jun 21;15:2619-2624. doi: 10.2147/OPTH.S320214. eCollection 2021. PMID 34188440